CLINICAL TRIAL: NCT02302534
Title: Pilot Study of Functional and Morphometric Brain Abnormalities Related to Adolescent Idiopathic Scoliosis (MOR-FO-SIA)
Acronym: MOR-FO-SIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO 2014 - JEL / MOR-FO-SIA
Record Dates: First submitted 2014-10-21; First posted 2014-11-27 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: scoliosis; MRI (Magnetic Resonance Imaging)
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Experimental): 2 groups with MRI :
  - 8 right thoracic AIS participants (Cobb angle between 20 and 40°)
  Interventions: Device: MRI
- controls subjects (Experimental): - 8 healthy controls (no clinical scoliosis)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a complex deformity with different curves. These different curves may be distinguished by different physiopathologic mechanisms.

Without fully convincing model of the emergence and development of AIS, their multifactorial nature seems evident. Several pathophysiological theories involving the central nervous system have been proposed: the AIS would be associated with disturbances of proprioceptive or sensory perception, and/or with integration of this information. This would result in an abnormal body image, responsible for sensorimotor asymmetry that may promote or cause the deformation.

The Main aim of this study is to find cortical and subcortical morphometric differences in the most common population of AIS (right thoracic AIS) compared to healthy adolescent control girls.

Secondary Objectives are to study the cerebral white matter of the same groups (fractional anisotropy in the main white matter tracts), and activation of sensorimotor neural networks (fMRI activation and functional brain connectivity).

Abnormalities of the studied parameters may be used as biomarkers for AIS diagnosis and classification.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 14 and 16 years old
* normal neurological examination
* right handed
* informed consent
* informed consent form signed by a parent or a holder of parental authority
* affiliated to medical insurance
* negative urine pregnancy test For patients (A-STD) : right thoracic scoliosis with a Cobb angle between 20 and 40° For healthy volunteers (A-N) : no clinical scoliosis

Exclusion Criteria:

* pregnant or lactating woman
* antecedents of cranial trauma or cranial intervention, of migraine, of spinal trauma, of scoliosis intervention
* no idiopathic scoliosis
* contraindications to MRI
* patient with a legal protection measure

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Variation in regional cortical and subcortical volume, as measured by MRI | One day

SECONDARY OUTCOMES:
Variation in fractional anisotropy in the main white matter tracts, as measured by MRI | one day
Variation in activation of sensorimotor neural networks, as measured by MRI | one day

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Edouard LORET, MD, Principal Investigator — University Hospital of Tours
Locations (1):
- University Hospital of Tours, Tours, France